CLINICAL TRIAL: NCT06306092
Title: Promoting Teenage Sleep - for Better Mental Health and School Performance
Brief Title: Promoting Teenage Sleep for Improved Mental Health and School Performance
Acronym: TeenSleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kristianstad University (Other)
Collaborators: Karolinska Institutet (Other); Örebro University, Sweden (Other); Academic Primary Health Care Centre, Region Stockholm (Unknown)
Responsible Party: Principal Investigator, Pernilla Garmy, Professor, Kristianstad University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-02885-01
Record Dates: First submitted 2023-11-30; First posted 2024-03-12 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Mental Health Issue; Insomnia; Depression; Anxiety; Daytime Sleepiness; Wellness, Psychological
Keywords: Sleep; Mental health; Adolescents; School-based intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Anxiety Disorders; Disorders of Excessive Somnolence; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "Sleep on Schedule" - sleep education at school (Experimental): The sleep training includes five lessons during school hours, and will be held by school staff (teachers, school nurses and school counsellors). The teaching consists of sleep education (sleep knowledge and good sleep routines), time management (e.g., planning homework without distraction, planning other activities, quiet time before bedtime), information to guardians, and discussions with peers in the classroom (e.g., rules regarding evening interaction via electronic media). Homework/exercises and behavioral experiments are also included. Data collection takes place in connection with the first and last lesson of Sleep on Schedule.
  Interventions: Behavioral: Sleep on Schedule
- "TechRest" - reduction of electronic media use before bedtime (Experimental): This intervention has been tested in Australia with a small sample of teenagers, and it was associated with promising effects. The data collection consists of a digital questionnaire regarding sleep habits, insomnia, motivation, physical and mental health, and electronic media use; a selection of students will use the actigraph for a week. After the first week, the participants will be instructed to stop using screens 1 hour before their usual bedtime. After one week has passed, participants in the Technology restriction intervention will be asked to complete the previously mentioned questionnaires as well as questions about the intervention itself: its applicability, compliance, and whether or not they will continue to limit their screen time before bedtime. One year after the intervention, they will be asked to complete the same questionnaire as at baseline. A selection of students will also wear a wrist actigraph.
  Interventions: Behavioral: Technology restriction
- Control (No Intervention): School as usual

INTERVENTIONS:
Behavioral: Sleep on Schedule — Sleep education at school
  Arms: "Sleep on Schedule" - sleep education at school
Behavioral: Technology restriction — Reduction of electronic media use before bedtime
  Arms: "TechRest" - reduction of electronic media use before bedtime

SUMMARY:
The overall aim of this project is to evaluate the effectiveness of two school-based programs that have the potential to promote adolescent sleep and prevent future depressive symptoms. The programs will be offered to students aged 13-19 at Swedish high schools and upper secondary schools at the classroom level. The students will be compared to teaching as usual (control group).

DETAILED DESCRIPTION:
Sleep problems are common among young people and there are connections between sleep problems and mental health, concentration problems, and lower grades. Over time (historically since the 80's), teenagers sleep less and less and too little, which affects mental health and school performance in the short term. Long-term lack of sleep increases the risk of leaving school with failed grades and of having long-term health problems. It is therefore important to break this trend.

A challenge in existing preventive sleep programs is to motivate young people to change their sleep habits. Just like adults, teenagers have many activities that demand their time. It can therefore be difficult to balance sleep with schoolwork, exercise, etc. Young people need knowledge about sleep to gain an understanding of how it can affect their mood and ability to cope with school. The reasons for the lack of sleep among young people are multifold: the 24-hour society and easily accessible entertainment/society via technology use, puberty-related changes in the circadian rhythm, and stress about the future. The school has a clear responsibility for the students' knowledge and understanding of the importance of lifestyle for health as well as for supporting the students in orienting themselves in society. The school is therefore a natural arena to reach out to teenagers because most young people are there, and the school health department can offer health-promotion initiatives.

The overall aim of this project is to evaluate the effectiveness of two school-based programs that have the potential to promote adolescent sleep and prevent future depressive symptoms. The programs will be offered to students aged 13-19 at Swedish high schools and upper secondary schools at the classroom level. The students will be compared to teaching as usual (control group).

Sleep on schedule is a program (5 lessons over 5 weeks) that integrates sleep knowledge and skill training to promote good sleep routines. Technology restriction is a program (2 lessons over 2 weeks) that targets mobile phone use at bedtime. Both programs have shown good results (up to 20 minutes more sleep on school days). The current goal was to test the effects of the programs on young people in a Swedish context to investigate if they can affect teenagers' sleep and mental health.

The study design is a cluster-randomized study where schools are randomized to either 1) Sleep on schedule, 2) Technology restriction, or 3) Control group (no intervention). All schools will be informed of the results and receive training in the program that proves to be most effective at the end of the project, if desired. The intervention is aimed at students aged 13-19. We want to involve large parts of the school's staff and avoid that knowledge and responsibility resting on a few members of staff. The program will be delivered by teachers or school health professionals (e.g., school counsellor, school nurse).

The interventions will directly benefit young people because sleep problems are a risk factor for mental illness and worse school performance. Sleep on schedule and restricting use of technology are important life skills and strategies that can help young people manage their everyday lives both now and in the future. The study offers benefits to the students in the intervention group in that they can learn strategies for preventive purposes regarding sleep before clinical problems arise. The participants will also have their voices heard on the subject.

ELIGIBILITY:
Inclusion Criteria:

Students in Swedish high schools and upper secondary schools.

Exclusion Criteria:

-

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3000 (Estimated)
Dates: Start 2024-08-17 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Change in sleep duration, hours and minutes | Baseline, 3 month, 1 year
  Self reported average time for sleep onset, time awake during the night and time for wakening in the morning, school days and weekends

SECONDARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale scores | Baseline, 3 month, 1 year
  Hospital Anxiety and Depression Scale measures anxiety and depression with 7 items for anxiety (range 0-21, higher scores mean worse outcome) and 7 items measure depression (range 0-21, higher scores mean worse outcome).
Change in Adolescent Sleep Hygiene Scale scores | Baseline, 3 month, 1 year
  Adolescent Sleep Hygiene Scale measures sleep habits, range 10-60, higher scores mean worse outcome.
Change in Insomnia Severity Index score | Baseline, 3 month, 1 year
  The Insomnia Severity Index (ISI) is a 7-item scale that asesses the severity of sleep disturbance, how much sleep disturbance interferes with daily life and functioning, the noticeability of these impairments to others, worry and distress resulting from sleep disturbance, and general sleep satisfaction/dissatisfaction. Responses are provided on a Likert-scale (0-4). The total score ranges from 0 to 28, and higher scores indicate more severe problems
Change in EuroQol Visual Analog Scale (EQ VAS) score | Baseline, 3 month, 1 year
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Change in CHU9D Child Health Utility 9D (CHU9D) scores | Baseline, 3 month, 1 year
  The CHU9D is a paediatric generic preference-based measure of health-related quality of life suitable for 7 to 17 year olds. It consists of a short questionnaire and a set of preference weights using general population values. The questionnaire has 9 questions with 5 response levels per question and is self-completed by the child. Range 9-45, higher scores mean worse outcome.
Change in Sleep knowledge | Baseline, 3 month, 1 year
  Sleep knowledge is measured with 9 questions, range 0-9, higher scores mean better sleep knowledge.
Change in electronic media use | Baseline, 3 month, 1 year
  Electronic media use is measured with 3 questions, range 3-12, higher scores mean more bedtime elecronic media use.
Change in sleep habits | Baseline, 3 month, 1 year
  Sleep habits regarding school days and weekends are measured with 10 questions.
Change in meta-cognitions | Baseline, 3 month, 1 year
  The Meta-Cognitions Questionnaire for Adolescents (MCQ-A) measures beliefs about worry and intrusive thoughts in adolescents aged between 13 and 17 year. Range 30-120, higher scores mean worse outcome.
Change in motivation | Baseline, 3 month, 1 year
  The Academic Self-Regulation Questionnaire (SRQ-A) - Intrinsic motivation subscale Why I do things measuer motivation. Range 7-28, higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Annika Norell, PhD, Principal Investigator — Örebro University, Sweden; Christina Sandlund, PhD, Principal Investigator — Karolinska Institutet; Pernilla Garmy, PhD, Principal Investigator — Kristianstad University; Serena Bauducco, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Kristianstad University, Kristianstad, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact pernilla.garmy@hkr.se
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 2030-2035

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT06306092/Prot_SAP_000.pdf